CLINICAL TRIAL: NCT05311904
Title: Observatory of the Efficacy and Safety of Vaccination Against SARS-CoV-2 in Neuromuscular Patients
Brief Title: Efficacy and Safety of Vaccination Against COVID-19 in Neuromuscular Patients
Acronym: VA-C-NEMUS
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2020/68
Record Dates: First submitted 2021-03-31; First posted 2022-04-05 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Neuromuscular Diseases
Keywords: COVID-19; vaccination; safety
MeSH Terms: conditions — Neuromuscular Diseases; COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — 1 initial questionnaire and 1 monthly follow-up questionnaire for 11 months

SUMMARY:
The frequency of severe forms of COVID-19 is higher in people with neuromuscular disease and in severe cases and long hospital stays, the disability of some neuromuscular patients may worsen due to prolonged bed rest . Finally, the symptoms of certain diseases such as myasthenia gravis can worsen after an infection such as COVID-19.

Thanks to an unprecedented research effort, vaccines are now available and others still in development. The first studies published in medical journals are reassuring about the efficacy and safety of these vaccines. However, they have been studied in the general population and we do not yet have specific information in neuromuscular patients.

This is the reason why the Va-C-NEMUS observatory was launched.

DETAILED DESCRIPTION:
Prevention of COVID-19 in neuromuscular patients is therefore fundamental and vaccination is eagerly awaited by patients and their healthcare teams. An unprecedented research effort has made it possible to create vaccines in a very short time when no vaccine directed against a coronavirus has existed until now. Some of these vaccines are based on proven technologies while others such as RNA vaccines are very innovative. The results of the phase III studies of 3 of them have just been published (Pfizer/BioNTech, Moderna and Astra-Zeneca). Among them, the Pfizer-BioNTech and Moderna vaccines have received authorization for use from the European Medicines Agency. The data on the individuals enrolled in these trials are still not very detailed. However, we already know that in the Pfizer/BioNTech trial, patients on immunosuppressants were excluded. For the Astra-Zeneca vaccine, the publication combines data from 4 different trials. In two of them the patients had to be in "good health". In any case, we do not know the pathologies presented by patients outside the usual risk factors for the severe form of COVID-19 (age, obesity, cardiovascular diseases, respiratory diseases). No data on neuromuscular patients are currently known. The vaccination campaign began in France in January 2021. The first neuromuscular patients should be vaccinated soon depending on their comorbidities, but many questions arise in these patients both in terms of safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with one of the following neuromuscular diseases:

   * Autoimmune myasthenia gravis, Lambert-Eaton syndrome
   * Congenital myasthenic syndromes
   * Myositis
   * Inflammatory neuropathies
   * Hereditary neuropathies (Charcot-Marie-Tooth disease, etc.)
   * Amyloid neuropathies
   * Spinal atrophies
   * Myotonic dystrophies type 1 (Steinert disease) and 2 (PROMM)
   * Duchenne and Becker muscular dystrophies
   * Muscular dystrophies of the girdles
   * Pump disease
   * Congenital myopathies
   * Congenital muscular dystrophies
   * Metabolic myopathies
   * Other myopathies with confirmed genetic diagnosis
2. Patient over 18 years old
3. Patient having understood that the follow-up of a possible side effect of the vaccination or of a COVID-19 must be carried out by his usual doctor (s) and not by the observatory team Va-C-NEMUS
4. Patients having been informed of the study and having expressed their agreement

Exclusion Criteria:

1. Patient under legal protection, curatorship or tutorship

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a neuromuscular disease
Sampling Method: Non-Probability Sample
Enrollment: 1388 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
the frequency of serious adverse reactions (SAEs) | at 1 month after the end of the vaccination against SARS-CoV-2 (after the 2nd injection for the majority of vaccines).
  the frequency of serious adverse reactions (SAEs) in the population of neuromuscular patients vaccinated against COVID19 Serious adverse reaction or event (Article R1123-46 of the Public Health Code and ICH-E2B guideline)
  Any adverse reaction or event that:
  * results in death,
  * endangers the life of the participant,
  * requires hospitalisation or prolongation of hospitalisation,
  * causes an inability or significant or long-term disability,
  * results in an abnormality or congenital malformation,
  * or any event considered to be medically serious, and with respect to the drug, regardless of the dose administered. The expression "life-threatening" is reserved for an immediate life threat at the time of the adverse event.
the frequency of unexpected adverse reactions (SUSARs) | at 1 month after the end of the vaccination against SARS-CoV-2 (after the 2nd injection for the majority of vaccines).
  Unexpected adverse event or suspected adverse reaction refers to an event or reaction that is not listed in the investigator's brochure or is not listed at the specificity or severity that has been observed; or, if an investigator's brochure is not required or available, is not consistent with the risk information

SECONDARY OUTCOMES:
vaccination's global safety : Frequency of Adverse Effects (AEs) | at 1 month after the end of the vaccination against SARS-CoV-2 (after the 2nd injection for the majority of vaccines).
  Frequency of Adverse Effects (AEs) in the population of neuromuscular patients vaccinated against COVID19
Risk of worsening autoimmune myasthenia gravis after vaccination | at 1 month after the end of the vaccination against SARS-CoV-2 (after the 2nd injection for the majority of vaccines).
  Myasthenia Gravis Foundation of America classification
Frequency of worsening of the autonomy of the patients evaluated with the MG-ADL | at 1 month after the end of the vaccination against SARS-CoV-2 (after the 2nd injection for the majority of vaccines).
  Frequency of worsening of the MG-ADL activity score by more than 2 points between the week before vaccination and the week following vaccination will be evaluated The Myasthenia Gravis-specific Activities of Daily Living scale consists of the assessment of 8 parameters: speaking, chewing, swallowing, breathing, self-care activities (brushing the teeth or combing the hair), simple physical activities (getting up from a chair), double vision and eye lid dropping. Each parameter is subjected to assessment depending on the degree of symptoms intensification, awarding points from 0 to 3 points. The maximum number a patient may receive is 24 points. The higher the score of points, the bigger limitations of the patient in everyday life activities caused by intensification of myasthenia gravis (Wolfe GI, Herbelin L, Nations SP, Foster B, Bryan WW, Barohn RJ. Myasthenia gravis activities of daily living profile. Neurology 1999;52:1487-1489.)
Frequency of hospitalizations for myasthenic crisis | at 1 month after the end of the vaccination against SARS-CoV-2 (after the 2nd injection for the majority of vaccines).
  Frequency of hospitalizations for myasthenic crisis in the month following vaccination
effectiveness of the vaccination | at least 7 days after the end of the vaccination against SARS-CoV-2 (after the 2nd injection for the majority of vaccines).
  Frequency of COVID-19 cases confirmed by a PCR test or an antigen test
effectiveness of the vaccination | at 1 month after the end of the vaccination against SARS-CoV-2 (after the 2nd injection for the majority of vaccines).
  Frequency of COVID-19 cases confirmed by a PCR test or an antigen test occurring
effectiveness of the vaccination | at 2 months after the end of the vaccination against SARS-CoV-2 (after the 2nd injection for the majority of vaccines).
  Frequency of COVID-19 cases confirmed by a PCR test or an antigen test occurring
effectiveness of the vaccination | at 3 months after the end of the vaccination against SARS-CoV-2 (after the 2nd injection for the majority of vaccines).
  Frequency of COVID-19 cases confirmed by a PCR test or an antigen test occurring
effectiveness of the vaccination | at 4 months after the end of the vaccination against SARS-CoV-2 (after the 2nd injection for the majority of vaccines).
  Frequency of COVID-19 cases confirmed by a PCR test or an antigen test occurring
effectiveness of the vaccination | at 5 months after the end of the vaccination against SARS-CoV-2 (after the 2nd injection for the majority of vaccines).
  Frequency of COVID-19 cases confirmed by a PCR test or an antigen test occurring
effectiveness of the vaccination | at 6 months after the end of the vaccination against SARS-CoV-2 (after the 2nd injection for the majority of vaccines).
  Frequency of COVID-19 cases confirmed by a PCR test or an antigen test occurring
the frequency of serious adverse reactions (SAEs) at 2 months | at 2 months after the end of the vaccination against SARS-CoV-2 (after the 2nd injection for the majority of vaccines).
  the frequency of serious adverse reactions (SAEs) in the population of neuromuscular patients vaccinated against COVID19 Serious adverse reaction or event (Article R1123-46 of the Public Health Code and ICH-E2B guideline)
  Any adverse reaction or event that:
  * results in death,
  * endangers the life of the participant,
  * requires hospitalisation or prolongation of hospitalisation,
  * causes an inability or significant or long-term disability,
  * results in an abnormality or congenital malformation,
  * or any event considered to be medically serious, and with respect to the drug, regardless of the dose administered. The expression "life-threatening" is reserved for an immediate life threat at the time of the adverse event.
the frequency of serious adverse reactions (SAEs) at 3 months | at 3 months after the end of the vaccination against SARS-CoV-2 (after the 2nd injection for the majority of vaccines).
  the frequency of serious adverse reactions (SAEs) in the population of neuromuscular patients vaccinated against COVID19 Serious adverse reaction or event (Article R1123-46 of the Public Health Code and ICH-E2B guideline)
  Any adverse reaction or event that:
  * results in death,
  * endangers the life of the participant,
  * requires hospitalisation or prolongation of hospitalisation,
  * causes an inability or significant or long-term disability,
  * results in an abnormality or congenital malformation,
  * or any event considered to be medically serious, and with respect to the drug, regardless of the dose administered. The expression "life-threatening" is reserved for an immediate life threat at the time of the adverse event.
the frequency of serious adverse reactions (SAEs) at 4 months | at 4 months after the end of the vaccination against SARS-CoV-2 (after the 2nd injection for the majority of vaccines).
  the frequency of serious adverse reactions (SAEs) in the population of neuromuscular patients vaccinated against COVID19 Serious adverse reaction or event (Article R1123-46 of the Public Health Code and ICH-E2B guideline)
  Any adverse reaction or event that:
  * results in death,
  * endangers the life of the participant,
  * requires hospitalisation or prolongation of hospitalisation,
  * causes an inability or significant or long-term disability,
  * results in an abnormality or congenital malformation,
  * or any event considered to be medically serious, and with respect to the drug, regardless of the dose administered. The expression "life-threatening" is reserved for an immediate life threat at the time of the adverse event.
the frequency of serious adverse reactions (SAEs) at 5 months | at 5 months after the end of the vaccination against SARS-CoV-2 (after the 2nd injection for the majority of vaccines).
  the frequency of serious adverse reactions (SAEs) in the population of neuromuscular patients vaccinated against COVID19 Serious adverse reaction or event (Article R1123-46 of the Public Health Code and ICH-E2B guideline)
  Any adverse reaction or event that:
  * results in death,
  * endangers the life of the participant,
  * requires hospitalisation or prolongation of hospitalisation,
  * causes an inability or significant or long-term disability,
  * results in an abnormality or congenital malformation,
  * or any event considered to be medically serious, and with respect to the drug, regardless of the dose administered. The expression "life-threatening" is reserved for an immediate life threat at the time of the adverse event.
the frequency of serious adverse reactions (SAEs) at 6 months | at 6 months after the end of the vaccination against SARS-CoV-2 (after the 2nd injection for the majority of vaccines).
  the frequency of serious adverse reactions (SAEs) in the population of neuromuscular patients vaccinated against COVID19 Serious adverse reaction or event (Article R1123-46 of the Public Health Code and ICH-E2B guideline)
  Any adverse reaction or event that:
  * results in death,
  * endangers the life of the participant,
  * requires hospitalisation or prolongation of hospitalisation,
  * causes an inability or significant or long-term disability,
  * results in an abnormality or congenital malformation,
  * or any event considered to be medically serious, and with respect to the drug, regardless of the dose administered. The expression "life-threatening" is reserved for an immediate life threat at the time of the adverse event.
the frequency of unexpected adverse reactions (SUSARs) at 2 months | at 2 months after the end of the vaccination against SARS-CoV-2 (after the 2nd injection for the majority of vaccines).
  Unexpected adverse event or suspected adverse reaction refers to an event or reaction that is not listed in the investigator's brochure or is not listed at the specificity or severity that has been observed; or, if an investigator's brochure is not required or available, is not consistent with the risk information
the frequency of unexpected adverse reactions (SUSARs) at 3 months | at 3 months after the end of the vaccination against SARS-CoV-2 (after the 2nd injection for the majority of vaccines).
  Unexpected adverse event or suspected adverse reaction refers to an event or reaction that is not listed in the investigator's brochure or is not listed at the specificity or severity that has been observed; or, if an investigator's brochure is not required or available, is not consistent with the risk information
the frequency of unexpected adverse reactions (SUSARs) at 4 months | at 4 months after the end of the vaccination against SARS-CoV-2 (after the 2nd injection for the majority of vaccines).
  Unexpected adverse event or suspected adverse reaction refers to an event or reaction that is not listed in the investigator's brochure or is not listed at the specificity or severity that has been observed; or, if an investigator's brochure is not required or available, is not consistent with the risk information
the frequency of unexepected adverse reactions (SUSARs) at 5 months | at 5 months after the end of the vaccination against SARS-CoV-2 (after the 2nd injection for the majority of vaccines).
  Unexpected adverse event or suspected adverse reaction refers to an event or reaction that is not listed in the investigator's brochure or is not listed at the specificity or severity that has been observed; or, if an investigator's brochure is not required or available, is not consistent with the risk information
the frequency of unexpected adverse reactions (SUSARs) at 6 months | at 6 months after the end of the vaccination against SARS-CoV-2 (after the 2nd injection for the majority of vaccines).
  Unexpected adverse event or suspected adverse reaction refers to an event or reaction that is not listed in the investigator's brochure or is not listed at the specificity or severity that has been observed; or, if an investigator's brochure is not required or available, is not consistent with the risk information

CONTACTS AND LOCATIONS:
Overall Officials: Guilhem SOLE, MD, Principal Investigator — Université Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France